CLINICAL TRIAL: NCT02908841
Title: Surgicel Snow in Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danbury Hospital (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Principal Investigator, Joann Petrini, PhD, MPH, Director, Clinical Outcomes and Health Services Research, Danbury Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-02-37-337
Record Dates: First submitted 2016-09-07; First posted 2016-09-21 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Laparoscopic Hysterectomy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): 30 patients randomized to the control group and will receive standard of care. Control patients will be managed with direct compression with gauze pads or laparotomy pads for four minutes. If hemostasis is not achieved by compression after four minutes, the source and rate of bleeding will be reevaluated and management will be determined by the surgeon. If the surgeon uses SurgicelSnow to achieve hemostasis at some point after 4 minutes, the patient will be included in the control group, but the data will be and flagged for the analysis. If failure of hemostasis at 4 minutes with an estimated loss of ≥25 cc/min, patient will be managed as per judgment of surgeon. Persistent bleeding at the 10 minute observation point will be treated as per the surgeon's judgment.
  Interventions: Other: Standard of Care
- Treatment (Other): 30 patients randomized to the treatment group will receive Surgicel Snow. For patients with qualifying bleeding (rated on initial evaluation as at least "mild") who have been randomized to receive Surgicel Snow, a single thin layer of dry Surgicel Snow will be applied over the area of bleeding and positioned firmly in direct contact to the areas of bleeding with blunt surgical instruments. Surgicel Snow will be left in the cavity to be absorbed. Dry gauze will not be placed over the material. No adjuncts will be added to the enhance hemostasis, but patients with small arteriolar bleeding will have pressure maintained on the bleeding site for 60 seconds. Hemostatic failure at 4 minutes will be reassessed for rate of blood loss and if the rate of loss is estimated at less than 25 cc per minute, additional observations will be made at 7 and 10 minutes.
  Interventions: Device: Surgicel Snow

INTERVENTIONS:
Device: Surgicel Snow
  Arms: Treatment
Other: Standard of Care
  Arms: Control

SUMMARY:
Surgicel Snow is an FDA approved topical hemostatic agent for use during surgical procedures. Like the other mechanical agents, Surgicel Snow forms a physical barrier that blocks blood flow while providing a large surface area for the rapid formation of a fibrin clot. As a mechanical agent derived from oxidized regenerated cellulose, Surgicel Snow shares with other mechanical hemostatic agents, the benefits of a favorable risk profile. This study would examine the efficacy of Surgicel Snow vs. direct compression in the control of capillary, venous, and small arterial hemorrhage when ligation or other conventional methods of control are impractical or ineffective in patients undergoing laparoscopic or robotic assisted laparoscopic hysterectomy. The intraoperative inclusion bleeding characteristics are minimal and mild retroperitoneal bleeding and moderate retroperitoneal bleeding that has been adequately reduced by standard surgical methods. 60 patients will be recruited for this study, all of which will be scheduled for hysterectomy at Western Connecticut Health Network (Norwalk Hospital and Danbury Hospital) under the direction of Dr. Thomas Rutherford, Dr. John Garofalo, and Dr. Robert Samuelson. The investigators will randomize 30 patients to the treatment group and 30 patients to the control group. Participants may continue all regular medications before and during the study. The consent process will be incorporated into the last pre-operative office visit. The health risks associated with use of Surgicel Snow may be less, the same or more than direct pressure alone. Surgicel Snow is generally used for minimal to mild bleeding from specific or widespread area; however, its effectiveness compared to direct pressure is unknown for a hysterectomy surgery.

DETAILED DESCRIPTION:
Topical hemostatic agents have been introduced as adjunct therapies to standard surgical techniques in the management of intraoperative bleeding. They are particularly useful in widespread non-anatomic bleeding or bleeding involving sensitive tissues. Topical hemostatic agents can be classified into four broad categories based on function: mechanical agents, biologic agents, flowable sealants, and fibrin sealants. Mechanical agents derived from oxidized regenerated cellulose forms a physical barrier to block blood flow, while providing a large surface area for rapid fibrin clot formation. The benefit of this mechanical agent includes a favorable risk profile. They are inexpensive, rapidly absorbed, rarely induces a local inflammatory response or fibrosis, and no reported potential for inducing immunological response or anaphylaxis.

In current literature, oxidized regenerated cellulose has been shown to reduce the length of stay and resource utilization in cardiovascular and neurologic procedures. Although these agents are being used with increasing frequency, there is a paucity of evidence to support a similar benefit in gynecologic surgery with the exception of a small number of studies on myomectomy and ovarian surgery. Although it is known that all of the agents presently approved by the FDA are capable of shortening the bleeding time associated with surgical incisions, there are limited studies to show comparative efficacy or clinical impact with respect to estimated blood loss in the retroperitoneal space. The results of extensive bleeding in the retroperitoneal spaces include significant blood loss with dissection along the extraperitoneal fascial planes, as well as intraperitoneal collection, hematoma, and abscess. Patients with postoperative pelvic collections may present with symptoms of fever, rectal pain, or lower abdominal pain. Treatment often requires IR (interventional radiology) drainage and readmission for inpatient parenteral antibiotic therapy. The initial approach to hemostasis in the pelvis depends on the nature of bleeding encountered. When bleeding is encountered during pelvic dissection, evaluation of the extent and sources of bleeding, as well as its anatomic location and proximity to vital structures are the first requirements. The process of evaluating bleeding requires inspection of the bleeding sites augmented by irrigation, suctioning, and blotting with gauze. Through this process, the rate (minimal, mild, moderate, and severe) , distribution (local vs. diffuse), anatomic site (i.e., if in close proximity to vital structures), and source of blood loss (small arterial, venous or capillary) is ascertained.

In this study, investigators would examine the efficacy of Surgicel Snow, a topical mechanical hemostatic agent, versus direct compression in the control of capillary, venous, and small arterial hemorrhage when ligation or other conventional methods of control are impractical or ineffective in patients undergoing laparoscopic or robotic assisted laparoscopic hysterectomy.

Primary Outcomes:

* Time to hemostasis
* Failure to achieve hemostasis

Secondary Outcomes:

* Total intraoperative time
* Intraoperative blood loss

ELIGIBILITY:
Inclusion criteria:

1. Women ≥18 years of age
2. Women scheduled for standard multiport laparoscopic, single site laparoscopic, and robotic assisted laparoscopic hysterectomy.
3. Sites of surgery include Norwalk Hospital and Danbury Hospital.
4. Indication for surgery includes benign, complex benign, and malignant conditions.
5. Signed informed consent

Exclusion criteria:

1. Vaginal hysterectomy or open abdominal hysterectomy;
2. Congenital or acquired coagulation disorder including recent (within 7 days of surgery) therapeutic anticoagulation or use agents affecting platelet function, other than low dose aspirin. (Preoperative prophylactic heparin is not an exclusion criterion.)
3. Hysterectomy at the time of sacrocolpopexy.
4. Ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joann Petrini, PhD, Study Chair — Nuvance Health
Locations (3):
- United States (3):
  - Danbury Hospital, Danbury, Connecticut
  - Physicians for Women's Health, Norwalk, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spangler D, Rothenburger S, Nguyen K, Jampani H, Weiss S, Bhende S. In vitro antimicrobial activity of oxidized regenerated cellulose against antibiotic-resistant microorganisms. Surg Infect (Larchmt). 2003 Fall;4(3):255-62. doi: 10.1089/109629603322419599. PMID 14588160
- [Background] Martyn D, Kocharian R, Lim S, Meckley LM, Miyasato G, Prifti K, Rao Y, Riebman JB, Scaife JG, Soneji Y, Corral M. Reduction in hospital costs and resource consumption associated with the use of advanced topical hemostats during inpatient procedures. J Med Econ. 2015 Jun;18(6):474-81. doi: 10.3111/13696998.2015.1017503. Epub 2015 Mar 26. PMID 25728820
- [Background] Ata B, Turkgeldi E, Seyhan A, Urman B. Effect of hemostatic method on ovarian reserve following laparoscopic endometrioma excision; comparison of suture, hemostatic sealant, and bipolar dessication. A systematic review and meta-analysis. J Minim Invasive Gynecol. 2015 Mar-Apr;22(3):363-72. doi: 10.1016/j.jmig.2014.12.168. Epub 2015 Jan 5. PMID 25573183
- [Background] Santulli P, Marcellin L, Touboul C, Ballester M, Darai E, Rouzier R. Experience with TachoSil in obstetric and gynecologic surgery. Int J Gynaecol Obstet. 2011 May;113(2):112-5. doi: 10.1016/j.ijgo.2010.11.019. Epub 2011 Mar 30. PMID 21453918
- [Background] Angioli R, Muzii L, Montera R, Damiani P, Bellati F, Plotti F, Zullo MA, Oronzi I, Terranova C, Panici PB. Feasibility of the use of novel matrix hemostatic sealant (FloSeal) to achieve hemostasis during laparoscopic excision of endometrioma. J Minim Invasive Gynecol. 2009 Mar-Apr;16(2):153-6. doi: 10.1016/j.jmig.2008.11.007. Epub 2009 Jan 9. PMID 19138574
- [Background] Ribeiro SC, Reich H, Rosenberg J, Guglielminetti E, Vidali A. Laparoscopic myomectomy and pregnancy outcome in infertile patients. Fertil Steril. 1999 Mar;71(3):571-4. doi: 10.1016/s0015-0282(98)00483-x. PMID 10065802
- [Background] Raga F, Sanz-Cortes M, Bonilla F, Casan EM, Bonilla-Musoles F. Reducing blood loss at myomectomy with use of a gelatin-thrombin matrix hemostatic sealant. Fertil Steril. 2009 Jul;92(1):356-60. doi: 10.1016/j.fertnstert.2008.04.038. Epub 2009 May 6. PMID 19423098
- [Background] Angioli R, Plotti F, Ricciardi R, Terranova C, Zullo MA, Damiani P, Montera R, Guzzo F, Scaletta G, Muzii L. The use of novel hemostatic sealant (Tisseel) in laparoscopic myomectomy: a case-control study. Surg Endosc. 2012 Jul;26(7):2046-53. doi: 10.1007/s00464-012-2154-2. Epub 2012 Feb 1. PMID 22302534
- [Background] Shander A, Kaplan LJ, Harris MT, Gross I, Nagarsheth NP, Nemeth J, Ozawa S, Riley JB, Ashton M, Ferraris VA. Topical hemostatic therapy in surgery: bridging the knowledge and practice gap. J Am Coll Surg. 2014 Sep;219(3):570-9.e4. doi: 10.1016/j.jamcollsurg.2014.03.061. Epub 2014 Jun 2. No abstract available. PMID 25151345
- [Background] Wysham WZ, Roque DR, Soper JT. Use of topical hemostatic agents in gynecologic surgery. Obstet Gynecol Surv. 2014 Sep;69(9):557-63. doi: 10.1097/OGX.0000000000000106. PMID 25229825
- [Background] Parker WH, Wagner WH. Gynecologic surgery and the management of hemorrhage. Obstet Gynecol Clin North Am. 2010 Sep;37(3):427-36. doi: 10.1016/j.ogc.2010.05.003. PMID 20674784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 43 patients were enrolled in the study, 21 patients were excluded due to lack of intraoperative bleeding.
Groups:
- Control: 10 patients randomized to the control group and received standard of care. Control patients were managed with direct compression with gauze pads or laparotomy pads for four minutes. If hemostasis was not achieved by compression after four minutes, the source and rate of bleeding were reevaluated and management was determined by the surgeon. If the surgeon used SurgicelSnow to achieve hemostasis at some point after 4 minutes, the patient was included in the control group, but the data was flagged for the analysis. If failure of hemostasis at 4 minutes with an estimated loss of ≥25 cc/min, patient was managed as per judgment of surgeon. Persistent bleeding at the 10 minute observation point was treated as per the surgeon's judgment.
  Standard of Care
- Treatment: 12 patients randomized to the treatment group received Surgicel Snow. For patients with qualifying bleeding (rated on initial evaluation as at least "mild") who have been randomized to receive Surgicel Snow, a single thin layer of dry Surgicel Snow was applied over the area of bleeding and positioned firmly in direct contact to the areas of bleeding with blunt surgical instruments. Surgicel Snow was left in the cavity to be absorbed. Dry gauze was not placed over the material. No adjuncts was added to the enhance hemostasis, but patients with small arteriolar bleeding, pressure was maintained on the bleeding site for 60 seconds. Hemostatic failure at 4 minutes was reassessed for rate of blood loss and if the rate of loss was estimated at less than 25 cc per minute, additional observations were made at 7 and 10 minutes.
  Surgicel Snow
Period: Overall Study
Arm/Group | Control | Treatment
Started | 10 | 12
Completed | 6 | 12
Not Completed | 4 | 0
Not completed — Physician Decision | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Standard of Care
- Treatment: Surgicel Snow
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (8.6) | 45.4 (8.8) | 50.3 (10.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
BMI [Mean (Standard Deviation); unit: kilograms/metres2] | 33.9 (10.3) | 28.8 (4.1) | 30.5 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bleeding at Specified Time Intervals
Description: Because multiple factors other than retroperitoneal bleeding contribute to the total intraoperative bleed loss, the investigators believe that the intraoperative estimated blood loss is not a pure indicator of the efficacy of a topical hemostatic agent for control of retroperitoneal bleeding. Data from the specified time points (4 minutes, 7 minutes and 10 minutes) was combined to calculate an average bleeding event time for each subject.
Time Frame: 4 minutes, 7 minutes and 10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Treatment
Number analyzed (Participants) | 6 | 12
seconds | 485.7 (432.3) | 199.1 (72.8)

2. Secondary Outcome: Total Intraoperative Time
Description: Total intraoperative was collected from medical record.
Time Frame: up to 4 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Treatment
Number analyzed (Participants) | 6 | 12
minutes | 166.2 (37.4) | 236.2 (54.0)

3. Secondary Outcome: Rate of Intraoperative Blood Loss
Description: Intraoperative blood loss data was collected from medical record.
Time Frame: up to 4 hours
Measure: Mean (Standard Deviation); unit: cubic centimeter/minute
Arm/Group | Control | Treatment
Number analyzed (Participants) | 6 | 12
cubic centimeter/minute | 82.5 (50.4) | 214.1 (126.4)

4. Secondary Outcome: Blood Transfusion
Description: Blood transfusion details was collected from medical record.
Time Frame: up to 4 hours
Measure: Mean (Standard Deviation); unit: cubic centimetre
Arm/Group | Control | Treatment
Number analyzed (Participants) | 6 | 12
cubic centimetre | NA (NA) — no participants in the Control Arm/Group had transfusions | 172.2 (402.4)

5. Secondary Outcome: Total Postoperative Symptomatic Fluid Collection
Description: Postoperative symptomatic fluid collection data collected at 2 week and 6 week time period was obtained from medical record. Data from 2 week and 6 week time points was combined to calculate the total postoperative symptomatic fluid collection for each subject.
Time Frame: through study completion, an average of 6 weeks
Measure: Mean (Standard Deviation); unit: cc/weeks
Arm/Group | Control | Treatment
Number analyzed (Participants) | 6 | 12
cc/weeks | NA (NA) — no participants in the Control Arm/Group had postoperative symptomatic fluid discharge | NA (NA) — no participants in the Treatment Arm/Group had postoperative symptomatic fluid discharge

6. Secondary Outcome: Number of Participants With Postoperative Pelvic Abscess
Description: Postoperative pelvic abscess data was collected from medical record.
Time Frame: through study completion, an average of 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 6 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each subject from the time informed consent was signed until termination from the study, up to 6 weeks
Groups:
- Control: Subjects randomized to the control group and received standard of care.
- Treatment: Subjects randomized to the treatment group received Surgicel Snow.
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/10 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=10) | Treatment (N=12)
Bowel perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient required subsequent surgery to repair bowel perforation which occurred during surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT02908841/Prot_SAP_000.pdf